CLINICAL TRIAL: NCT00324974
Title: A Phase 3, Randomized, Multi-Center, Double-Blind, Placebo-Controlled, Parallel Group Study Assessing the Safety and Efficacy of Lansoprazole Microgranules Oral Suspension in Infants With Symptomatic Gastroesophageal Reflux
Brief Title: The Use of Lansoprazole to Treat Infants With Symptoms of Gastroesophageal Reflux
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP Clinical Sciences, Takeda Global Research & Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P-GI05-109; 2006-000957-23 (EudraCT Number); U1111-1114-2358 (Registry Identifier: WHO)
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2010-07

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal Reflux Disease; infant; lansoprazole oral suspension; PPI
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lansoprazole QD (Experimental)
  Interventions: Drug: Lansoprazole microgranules suspension
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lansoprazole microgranules suspension — Lansoprazole microgranules 0.2-0.3 mg/kg/day suspension, orally, once daily for up to 28 days for infants less than 10 weeks;
  Lansoprazole microgranules 1.0-1.5 mg/kg/day suspension, orally, once daily for up to 28 days for infants greater than 10 weeks.
  Arms: Lansoprazole QD
Drug: Placebo — Lansoprazole placebo-matching suspension, orally, once daily for up to 28 days.
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to assess the safety and efficacy of lansoprazole microgranules oral suspension, once daily (QD), in infants with gastroesophageal reflux symptoms during a 4-week treatment period.

DETAILED DESCRIPTION:
This study will be conducted by approximately 20 investigative sites in the U.S. and Poland. Participants who qualify will be randomized in equal proportions to receive either lansoprazole Pediatric Suspension (0.2-0.3 mg/kg/day in infants <10 weeks of age or 1.0-1.5 mg/kg/day in infants >10 weeks of age) or Placebo. This study consists of three periods: Pretreatment Period of 7-14 days, Double-Blind Treatment Period of 4 weeks (Dosing), and the Post-Treatment Period of 30 days (Follow-Up).

ELIGIBILITY:
Inclusion Criteria:

* At least 7 days post-surgery at the time of Screening (Study Visit 1) with no anticipated need for surgery during the study.
* Experiencing symptoms of gastroesophageal reflux disease (regurgitation, vomiting or "spitting up," fussing/irritability, feeding refusal, crying during feeding, arching back, poor weight gain, or extraesophageal manifestations) or endoscopy proven reflux disease.
* Must continue to have reflux symptoms during the Pretreatment Period despite reducing or eliminating exposure to tobacco smoke, using one positioning and feeding strategy the last 7 days as documented in the Daily Diary.
* The infant exhibited crying, fussing, or irritability during or within 1 hour of feeding in >25% of all feedings during the last 4 days of the Pretreatment Period as documented in the Daily Diary.

Exclusion Criteria:

* Body weight <2.0 kilogram at Dosing Day 1 of the Double-Blind Treatment Period.
* Unstable, congenital or acquired, clinically significant disease of any major organ system (cardiovascular, respiratory, renal, hepatic, metabolic, etc.), including suspected and/or documented culture-proven sepsis.
* Coexisting esophageal disease (e.g., eosinophilic esophagitis, viral, bacterial or fungal infection) or caustic or physiochemical trauma to the esophagus.
* Any congenital anomaly of the upper gastric intestinal tract that might interfere with gastrointestinal motility, pH, absorption, or active or known history of necrotizing enterocolitis that has been surgically corrected.
* Use of a proton pump inhibitor within 30 days prior to Dosing Day 1.
* Use of H2 Blockers (i.e. Zantac) within 7 days prior to Dosing Day 1.
* Allergy to proton pump inhibitors (i.e. Prilosec, Prevacid).
* Use of prokinetics (e.g., metoclopramide) unless on a stable dose for at least 3 days prior to entering the Pretreatment Period.
* Unable to obtain stable drug levels after continuous treatment with required drugs including theophylline derivatives, digoxin, phenytoin, phenobarbital, or carbamazepine within the 7 days prior to Dosing Day 1.
* Clinically Significant abnormalities in clinical laboratory values.

Ages: 1 Month to 11 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 162 (Actual)
Dates: Start 2006-06; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects in each treatment group responding to treatment with a reduction from baseline in the percentage and duration of crying/fussing/irritability episodes associated with feeding after 4 weeks of treatment. | Week 4
Safety Assessments | Baseline through week 8

SECONDARY OUTCOMES:
Global Symptom Assessment, as answered by Investigator and Parent/Guardian | Baseline through Week 8
Sensitivity analyses of the primary endpoint | Week 4
Additional Daily Diary-based symptom Assessments | At the end of the double-blind treatment period and 30 days after the last dose of study drug.
Indicators of Growth Parameters | During and at the end of the Double-blind treatment period and 30 days after the last dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (17):
- United States (9):
  - Tampa, Florida
  - Park Ridge, Illinois
  - Shreveport, Louisiana
  - Flint, Michigan
  - Omaha, Nebraska
  - Buffalo, New York
  - Cincinnati, Ohio
  - Youngstown, Ohio
  - Vienna, Virginia
- Poland (8):
  - Bialystok
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Rzeszów
  - Warsaw
  - Wroclaw

REFERENCES:
- [Result] Orenstein SR, Hassall E, Furmaga-Jablonska W, Atkinson S, Raanan M. Multicenter, double-blind, randomized, placebo-controlled trial assessing the efficacy and safety of proton pump inhibitor lansoprazole in infants with symptoms of gastroesophageal reflux disease. J Pediatr. 2009 Apr;154(4):514-520.e4. doi: 10.1016/j.jpeds.2008.09.054. Epub 2008 Dec 3. PMID 19054529